CLINICAL TRIAL: NCT07313566
Title: An Evidence-based Rehabilitation Pathway for Patients Undergoing Surgery for Lumbar Radicular Pain to Promote Return to Work: a Cluster Randomized Trial Comparison With Usual Care.
Brief Title: R³ Rehab Pathway Versus Usual Care After Lumbar Radicular Surgery
Acronym: R³
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Federal Knowledge Centre (KCE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S68181; KCE23-1473 (Other Grant/Funding Number: Belgian Health Care Knowledge Centre Trials Program (KCE trials))
Record Dates: First submitted 2025-11-24; First posted 2026-01-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Radiculopathy; Radicular Low Back Pain
Keywords: Lumbar radiculopathy; Return to work; Case manager; Cluster RCT; Rehabilitation; radicular pain
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: R³ Rehabilitation Pathway (Experimental): A structured evidence-based rehabilitation pathway, guided by a case manager, starting preoperatively to 1 year postoperatively, including prehabilitation, perioperative rehabilitation and postoperative rehabilitation, with emphasis on fear reduction by keeping activity restrictions minimal and relevant, eliminating bracing and on active guidance to work resumption.
  Interventions: Other: R³ Rehabilitation Pathway
- Control: usual care (No Intervention): Usual care, i.e. usual, variable rehabilitation care, which may vary between and within hospitals and may include no rehabilitation, monodisciplinary or multidisciplinary care, with highly variable advice to the patients

INTERVENTIONS:
Other: R³ Rehabilitation Pathway — A structured evidence-based rehabilitation pathway, guided by a case manager, starting preoperatively to 1 year postoperatively, including prehabilitation, perioperative rehabilitation and postoperative rehabilitation, with emphasis on fear reduction by keeping activity restrictions minimal and relevant, eliminating bracing and on active guidance to work resumption.
  Arms: Intervention: R³ Rehabilitation Pathway

SUMMARY:
The R³ trial is a multicentre cluster randomized controlled trial evaluating an evidence-based, person-centred rehabilitation pathway for patients undergoing lumbar surgery for radicular pain. The pathway includes structured pre-, peri-, and postoperative rehabilitation, early postoperative mobilization, case management, early return-to-work (RTW) guidance, and patient empowerment. Clusters (hospitals) are randomized to implement the R³ pathway (intervention) or continue usual care (control). The primary aim is to determine whether the R³ pathway reduces time to return to work compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Radicular pain (for ≥ 6 weeks prior to screening), with a clear indication for lumbar spinal surgery ((micro)discectomy, decompression and/or fusion), in accordance with the KCE guidelines (when evidence-based multimodal management has not improved pain or function and radiological findings are consistent with clinical symptoms)
* Employed (working or on sick leave for less than 1 year due to spinal pathology)
* Age 18 - 65 years
* Surgery is scheduled within a timeframe of five days to 2 months after the decision for surgery (4 months for fusion)
* For lumbar fusion surgery, the fusion should be restricted to one or two levels
* Able to provide written informed consent, implying that the participant is both physically and cognitively capable of understanding the study information and signing the consent form independently.

Exclusion Criteria:

Patients are not eligible for the trial in case of any of the following criteria:

* Lumbar surgery performed for malignant disease, spinal fracture, infectious spinal disease
* Insufficient knowledge of Dutch or French language to receive education in the recruiting center and to complete the questionnaires (consistent with the language spoken in the recruiting centre)
* Immediate surgery via emergency admission that precludes prehabilitation
* Revision fusion surgery
* Non-residency in Belgium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Time to Return To Work (RTW) | Assessed from surgery to 15 months postoperatively
  Time to return to work, defined as at least 50% of the contractional work time before surgery (with a sustainable return to work being defined as remaining actively working for three months following work resumption).
  Outcome type: Time-to-event (days) Range: 0 to 450 days Interpretation: Shorter time indicates a better outcome

SECONDARY OUTCOMES:
Disability | 3 months and 12 months postoperatively
  Disability scores assessed by the Oswestry Disability Index (ODI) at 3 months and 1 year postoperatively (key-secondary)
  Scale range: 0-100 points Interpretation: Higher scores indicate greater disability (worse outcome)
Percentage of patients returned to work | 4 weeks, 3 months and 1 year postoperatively
  Percentage of patients returned to work at 4 weeks, 3 months and 1 year postoperatively
  Scale range: 0-100% Interpretation: Higher percentages indicate a better outcome
Patient-centered functional status | 4 weeks, 3 months and 1 year postoperatively
  Patient-centered functional status assessed by the Patient-Specific Functional Scale (PSFS) at 4 weeks, 3 months and 1 year postoperatively
  Scale range: 0-10 per activity (mean score calculated) Interpretation: Higher scores indicate better functional ability
Back pain | 4 weeks, 3 months and 1 year postoperatively
  Back pain measured with the Numeric Rating Scale (NRS) at 4 weeks, 3 months and 1 year postoperatively
  Scale range: 0-10 0 = no pain 10 = worst imaginable pain Interpretation: Higher scores indicate more severe pain (worse outcome)
Leg pain | 4 weeks, 3 months and 1 year postoperatively
  Leg pain measured with the Numeric Rating Scale (NRS) at 4 weeks, 3 months and 1 year postoperatively
  Scale range: 0-10 0 = no pain 10 = worst imaginable pain Interpretation: Higher scores indicate more severe pain (worse outcome)
Health-related quality of life | 4 weeks, 3 months and 1 year postoperatively
  EuroQoL 5D (EQ5D-5L) for measuring health-related quality of life at 4 weeks, 3 months and 1 year postoperatively
  Index score range:
  From <0 (health states worse than death) to 1.0 (full health) Interpretation: Higher scores indicate better health-related quality of life
Work productivity | 4 weeks, 3 months and 1 year postoperatively
  Work productivity measured with the IMTA Productivity Cost Questionnaire (iPCQ) at 4 weeks, 3 months and 1 year postoperatively
  Scale: Multiple items assessing absenteeism and presenteeism Range: Item-specific (continuous variables expressed in days or hours) Interpretation: Higher productivity loss indicates a worse outcome
Analgesics use | 4 weeks, 3 months and 1 year postoperatively
  Analgesics use, quantified by the Medication Quantification Scale (MQS) at 4 weeks, 3 months and 1 year postoperatively
  Scale range: 0 to no predefined maximum (higher scores reflect greater medication burden) Interpretation: Higher scores indicate greater analgesic use (worse outcome)
Kinesiophobia | 4 weeks, 3 months and 1 year postoperatively
  Kinesiophobia measured by the Tampa Scale for Kinesiophobia (TSK) at 4 weeks, 3 months and 1 year postoperatively
  Scale range: 17-68 Interpretation: Higher scores indicate greater fear of movement (worse outcome)
Pain catastrophizing | 4 weeks, 3 months and 1 year postoperatively
  Pain catastrophizing measured by the Pain Catastrophizing Scale (PCS) at 4 weeks, 3 months and 1 year postoperatively
  Scale range: 0-52 Interpretation: Higher scores indicate greater pain catastrophizing (worse outcome)

CONTACTS AND LOCATIONS:
Locations (16):
- Belgium (16):
  - ZAS, Antwerp
  - AZ Sint Jan Brugge, Bruges
  - UZ Brussel, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Ziekenhuis Geel, Geel
  - ZOL Genk, Genk
  - Jessa Ziekenhuis, Hasselt
  - AZ Herentals, Herentals
  - Jan Yperman ziekenhuis, Ieper
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven
  - Heilig Hart Lier, Lier
  - AZ Sint Maarten Mechelen, Mechelen
  - CSPO, Ottignies
  - AZ Delta Roeselare, Roeselare
  - Centre Hospitalier de Wallonie Picarde, Tournai

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcomes will be shared, including demographic variables, surgical characteristics, pain scores, disability measures, quality-of-life outcomes, work-status variables, and follow-up assessments. No identifying data will be shared. Data will be provided in a fully anonymized format in accordance with GDPR and institutional data protection standards.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting documents will become available 12 months after publication of the primary results of the trial. Data will remain available for a minimum of 5 years after publication. Requests can be submitted at any time within this window. After 5 years, continued availability will depend on data storage capacity and institutional policies.
Access Criteria: Access will be granted to qualified researchers with a methodologically sound proposal aimed at scientific replication or secondary analyses related to postoperative rehabilitation or return-to-work after lumbar surgery. Requests must include a study protocol and data management plan. Following review and approval by the study team, data will be shared through a secure institutional platform under a data-sharing agreement. Only fully anonymized datasets and approved supporting documents will be accessible.